CLINICAL TRIAL: NCT06800612
Title: Observational Study Evaluating the Efficacy and Tolerability of Anticancer Drug Therapies Adopted for the Treatment of Gynecologic and Breast Cancers in Clinical Practice Compared with the Results of Registration Studies
Brief Title: Evaluating Efficacy and Tolerability of Anticancer Drug Therapies for the Treatment of Gynecologic and Breast Cancers
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: STRATEGIA
Record Dates: First submitted 2024-12-27; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Cancer Metastatic; Ovarian Cancer; Cervical Carcinoma; Endometrial Cancer
Keywords: observational; breast cancer; gynecologic cancer; ovarian cancer; cervical carcinoma; endometrial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- retrospective cohort: In this cohort data will be recorded retrospectively
  Interventions: Drug: Oncologic drugs administered for treatment of breast cancer; Drug: Oncologic drug administered for treatment of gynecologic cancer
- prospective cohort: In this cohort data will be recorded prospectively
  Interventions: Drug: Oncologic drugs administered for treatment of breast cancer; Drug: Oncologic drug administered for treatment of gynecologic cancer

INTERVENTIONS:
Drug: Oncologic drugs administered for treatment of breast cancer — Data on oncologic drugs administered for treatment of breast cancer will be recorded
Drug: Oncologic drug administered for treatment of gynecologic cancer — Data on oncologic drugs administered for treatment of gynecologic cancer will be recorded

SUMMARY:
retrospective/prospective observational study. Objective of the study is to evaluate the effect of drugs in terms of objective responses, disease-free survival (DFS), progression-free survival (PFS), overall survival (OS), and side effects compared with registry studies in the medical therapy of breast and gynecologic cancers.

DETAILED DESCRIPTION:
This is a single-center retrospective/prospective observational study. Objective of the study is to evaluate the effect of drugs in terms of objective responses, disease-free survival (DFS), progression-free survival (PFS), overall survival (OS), and side effects compared with registry studies in the medical therapy of breast and gynecologic cancers.

Regarding the prospective component of the study, it is clarified that therapy will be warranted by clinical practice regardless of study enrollment. Diagnostic investigations will also be conducted as per normal practice; enrollment in the study does not require additional examinations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed breast cancer or gynecological cancer, either early stage or metastatic;
* Patients who have received treatment for breast cancer or gynecologic cancer since January 2010;
* Any patient currently living and actually contactable must sign an informed consent to the study and processing of personal data.

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients treated for breast or gynecologic cancer from January 2010.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  To evaluate effect of drugs in terms of objective responses compared with registrational studies in medical therapy of breast and gynecological cancers: disease-free survival (DFS)

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  Effect of drugs in terms of objective responses compared with registrational studies in medical therapy of breast and gynecological cancers: progression-free survival (PFS)
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  Effect of drugs in terms of objective responses compared with registrational studies in medical therapy of breast and gynecological cancers: overall survival (OS)
Side effects | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  Effect of drugs in terms of objective responses compared with registrational studies in medical therapy of breast and gynecological cancers: side effects

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Zamagni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy